CLINICAL TRIAL: NCT00501098
Title: A Multicenter Phase II Study to Evaluate the Safety, Tolerability and Efficacy of Caspofungin as Prophylactic Treatment of Invasive Fungal Infections in Patients With Acute Leukemia Undergoing Induction Chemotherapy
Brief Title: Prophylaxis of Fungal Invasive Infections in Leukemia
Acronym: PROFIL-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Italy Leukemia Group (Other)
Responsible Party: Giuseppe Rossi, Spedali Civili di Brescia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2006-004432-70
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Invasive Pulmonary Aspergillosis
Keywords: Leukemia; Prophylaxis; Fungal Infections; Caspofungin
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Leukemia; Mycoses | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Patients will receive caspofungin, starting from the first day of induction chemotherapy for leukemia, as a single daily dose intravenously at the dosage of 70 mg q.d. and followed by 50 mg q.d. thereafter until documentation of complete hematologic remission after the first induction cycle or of leukemia persistence after one cycle of induction and one cycle of salvage chemotherapy.
  No stratification is planned.
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — Patients will receive caspofungin, starting from the first day of induction chemotherapy for leukemia, as a single daily dose intravenously at the dosage of 70 mg q.d. and followed by 50 mg q.d. thereafter until documentation of complete hematologic remission after the first induction cycle or of leukemia persistence after one cycle of induction and one cycle of salvage chemotherapy.
  No stratification is planned.

SUMMARY:
* To assess the overall clinical yield - in terms of efficacy and safety endpoints of adding caspofungin as prophylaxis of Invasive Pulmonary Aspergillosis in patients undergoing induction treatment for newly diagnosed acute leukemia
* To investigate the prognostic significance of Ptx3 at diagnosis and during the first chemotherapy cycle with respect to the development of IPA

DETAILED DESCRIPTION:
Invasive aspergillosis (IA), and particularly invasive pulmonary aspergillosis (IPA), is an important cause of morbidity and mortality in patients who are receiving chemotherapy for acute leukemia (AL), being the the most common invasive mycosis which develops in these patients. Proven invasive aspergillosis has been reported in 6,5% of patients with acute leukemia in a retrospective multicenter study (Pagano, Haematologica 2001) but that frequency may be underestimated, since definite diagnosis is difficult to obtain, particularly in leukemic patients.

When the recently developed, internationally recognized IFIGC/MSG/EORTC diagnostic criteria were retrospectively applied to a consecutive series of acute leukemia patients, the overall frequency of IPA was 25,3% (proven/probable 8,5%; possible 16,9%). Criteria for a diagnosis of IPA were fulfilled in 62,8% of pulmonary infiltrates developing in AL patients (proven/probable 17,1%; possible 45,7%). IPA developed both in AML and in ALL patients. Proven/probable IPA developed in 83% of cases during the first induction cycle (Borlenghi, EHA 2003). It may be estimated that such figures would be higher when patients would be followed prospectively and strictly monitored, particularly with GM antigenemia.

The mechanisms by which common colonizing agents like Aspergillus spp. can become invasive pathogens and cause severe tissue damage are only partially known. Recent experimental data in animal models raised the hypothesis that the long pentraxin Ptx3 may play an important role in resistance to selected microbial agents, in particular to Aspergillus fumigatus (Garlanda, Nature 2002).

Caspofungin is an echinocandin with potent antifungal activity against Aspergillus species. Its mechanism of action differs from that of the antifungal agents used so far, like amphotericin and azoles. It has proven effective and well tolerated and its use is therefore currently approved as salvage treatment in patients with invasive aspergillosis refractory to amphotericin, as well as for the empiric treatment of febrile neutropenia. Indeed it has been recently evaluated as empirical treatment in neutropenic patients with persistent fever of unknown origin and proved equally effective and better tolerated than liposomal amphotericin.

There are as yet no data on the use of caspofungin as primary prophylaxis in patients with acute leukaemia, a setting in which the lack of effective preventive treatments together with the generally favourable safety profile and efficacy of caspofungin makes it particularly attractive for investigation.

It can be hypothesized from the above data that the administration of caspofungin as prophylactic treatment of invasive aspergillosis should be safe and well tolerated by patient undergoing chemotherapy for acute leukemia at diagnosis.

It may reduce the high incidence of invasive pulmonary aspergillosis which characteristically develops during the first course of induction treatment, avoiding the direct morbidity and mortality of IPA and its negative impact on the treatment and prognosis of AL as well as the costs for IPA diagnosis and treatment.

The serum levels of the long pentraxin Ptx3 may have interpatient variability and may correlate with the subsequent development of invasive aspergillosis.

These facts led to the present multicenter, phase II, single arm, open study, performed by the Northern Italy Leukemia Group. There will be approximately 12 participating centers, which will enroll a total of 100 patients. Patients will receive caspofungin, starting from the first day of induction chemotherapy for leukemia, as a single daily dose intravenously at the dosage of 70 mg q.d. and followed by 50 mg q.d. thereafter until documentation of complete hematologic remission after the first induction cycle or of leukemia persistence after one cycle of induction and one cycle of salvage chemotherapy.

No stratification is planned. Patients will concurrently receive all the medications needed for the treatment of acute leukemia,according to the ongoing protocols of NILG for acute leukemia at diagnosis. The study period continues

The treatment will be stopped in the presence of any of the following conditions:

* Development of a severe adverse event or of any grade 3-4 toxicity attributable to caspofungin
* Development of proven/probable IPA No caspofungin dose reduction is planned. The dose of caspofungin will be adjusted when patients weight is over 80 kgs and in patients taking rifampin or other liver enzymes-inducing drugs.

ELIGIBILITY:
Inclusion Criteria:

* all patients with a diagnosis af acute leukemia who are enrolled in the clinical protocols of NILG for acute leukemia at diagnosis
* age > 18
* written informed consent

Exclusion Criteria:

* presence of signs or symptoms suspected of invasive fungal infection at enrollment
* history of allergy, hypersensitivity, or any serious reaction to echinocandin
* pregnancy or breast-feeding
* acute hepatitis or moderate/severe hepatic insufficiency of any cause;
* concomitant treatment with any systemic antifungal agent
* recent prior use of caspofungin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of probable/proven invasive aspergillosis

SECONDARY OUTCOMES:
Death rate The rate of overall serious drug related AEs Variation in Ptx3 levels between patients, and in each patient at different times, and their correlation with the development of Invasive Pulmonary Aspergillosis.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Rossi, MD, Principal Investigator — Spedali Civili di Brescia; Chiara Cattaneo, Principal Investigator — Spedali Civili di Brescia
Locations (8):
- Italy (8):
  - Dipartimento di Ematologia e Medicina Trasfusionale - Azienda Osp. Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - USC Ematologia Ospedali Riuniti di Bergamo, Bergamo, BG
  - Ematologia Centro TMO - Fondazione IRCSS Ospedale Maggiore, Milan, MI
  - Ematologia - TMO - Ospedale San Gerardo, Monza, MI
  - Ematologia 2 - Osp. Molinette San Giovanni Battista, Torino, TO
  - Medicina Interna I Ospedale di Circolo, Varese, VA
  - Divisione Ematologia Ospedale Umberto I, Mestre, VE
  - Divisione Ematologia Spedali Civili, Azienda Ospedaliera, Spedali Civili di Brescia, Brescia

REFERENCES:
- [Derived] Cattaneo C, Monte S, Algarotti A, Audisio E, Borlenghi E, Campiotti L, Cerqui E, Fanizza C, Giuliani R, Mico C, Rocconi R, Salvi A, Salvi F, Verga L, Levis A, Lambertenghi Deliliers G, Pogliani EM, Tognoni G, Rambaldi A, Rossi G. A randomized comparison of caspofungin versus antifungal prophylaxis according to investigator policy in acute leukaemia patients undergoing induction chemotherapy (PROFIL-C study). J Antimicrob Chemother. 2011 Sep;66(9):2140-5. doi: 10.1093/jac/dkr271. Epub 2011 Jul 5. PMID 21729932